CLINICAL TRIAL: NCT00031421
Title: A Follow-up Assessment of Subjects Who Received Ganciclovir (Dihydroxypropoxymethyl Guanine [DHPG]) During the Phase I/II Study to Evaluate the Safety and Efficacy of Ganciclovir Treatment for Congenital Cytomegalovirus (CMV) Infections
Brief Title: Neonatal CMV-Ganciclovir Follow-up Study
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Robert Johnson, HHS/NIAID/DMID
Other Study IDs: 01-489; CASG 108; N01AI30025C; N01AI30025 (NIH)
Record Dates: First submitted 2002-03-06; First posted 2002-03-07 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2008-07

CONDITIONS: Cytomegalovirus Infections
Keywords: CMV, cytomegalovirus, children, ganciclovir
MeSH Terms: conditions — Cytomegalovirus Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- 1: 16 received ganciclovir at 8 mg/kg/day in the previous study.
- 2: 31 received ganciclovir at 12 mg/kg/day in the previous study.

SUMMARY:
The purpose of this study is to document the developments associated with puberty and determine if any of the children who previously participated in another research study have been diagnosed with cancer. The previous study was a Collaborative Antiviral Study Group (CASG) protocol entitled "Evaluation of Ganciclovir (DHPG) for the Treatment of Symptomatic Congenital Cytomegalovirus Infections." One of the medications used in this study to treat cytomegalovirus (CMV), ganciclovir, has been known to cause cancer and affect the development of gonads (ovaries in females and testes in males) when administered to animals. Children, 9-14 years old, who participated in the previous research study, will participate in this study for 1 day. Subjects will be evaluated by an endocrinologist and will have the following procedures performed: a complete physical examination, a single blood sample collected, an x-ray of the left wrist.

DETAILED DESCRIPTION:
Ganciclovir has been shown to be carcinogenic, teratogenic, and gonadal toxic in animal models. Mice treated with ganciclovir experienced an increase in the incidence of tumors of the preputial gland (males), harderian gland (males), forestomach (males and females), ovaries (females), uterus (females), mammary gland (females), clitoral gland (females), vagina (females), and liver (females). While the preputial and clitoral glands, forestomach, and harderian glands of mice do not have human counterparts, ganciclovir is considered a potential carcinogen in humans. Animal data indicate that administration of ganciclovir causes inhibition of spermatogenesis and subsequent infertility, possibly due to inhibition of rapidly dividing cell populations including spermatogonia. In the animal models, these effects were reversible at lower doses and irreversible at higher doses. In both male and female mice, ganciclovir has been shown to cause decreased fertility. Gonadal toxicity in rats, mice, and dogs included testicular atrophy in males and, more variable, ovarian atrophy in females. There are no data in humans that demonstrate these effects following treatment with ganciclovir. This study seeks to formally establish the overall sexual development, cancer incidence, and pubertal status of those study subjects who previously received six weeks of ganciclovir as they now approach puberty. The original study was performed from 1986 to 1991, and therefore subjects who were enrolled are now nine to fourteen years of age.

ELIGIBILITY:
Inclusion Criteria:

Children who received ganciclovir during the earlier study ("Evaluation of Ganciclovir (DHPG) for the Treatment of Symptomatic Congenital Cytomegalovirus Infections), and if the parent or legal guardian signs an informed consent and the child signs an assent (where appropriate).

Exclusion Criteria:

Any individuals not previously enrolled in the CASG protocol titled "Evaluation of Ganciclovir (DHPG) for the Treatment of Symptomatic Congenital Cytomegalovirus Infections"

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children of both genders that previously enrolled in "Evaluation of Ganciclovir (DHPG) for the Treatment of Symptomatice Congenital Cytomegalovirus Infections."
Sampling Method: Probability Sample
Enrollment: 8
Dates: Start 2001-09; Study Completion 2005-11

PRIMARY OUTCOMES:
Sexual Development. | Analysis.
Pubertal Status. | Analysis.
Cancer Incidence. | Analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States